CLINICAL TRIAL: NCT02985099
Title: 1.2% Rosuvastatin Subgingivally Delivered In Treatment Of Chronic Periodontitis With Type 2 Diabetes Mellitus: A Placebo Controlled Clinical Trial
Brief Title: 1.2% Rosuvastatin Subgingivally Delivered In Chronic Periodontitis With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and Head, Dept of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014DK
Record Dates: First submitted 2016-12-04; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Periodontitis; Type2 Diabetes
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Rosuvastatin group (Active Comparator): Oral prophylaxis followed by 1.2% Rosuvastatin drug in gel form placed in intrabony defects
  Interventions: Drug: SRP plus Rosuvastatin gel
- Placebo group (Placebo Comparator): Oral prophylaxis followed by placebo gel placement in intrabony defects
  Interventions: Drug: SRP plus placebo gel

INTERVENTIONS:
Drug: SRP plus Rosuvastatin gel — SRP followed by 1.2% Rosuvastatin placement into intrabony defect
  Arms: Rosuvastatin group
Drug: SRP plus placebo gel — SRP followed by placebo gel placement into intrabony defect
  Arms: Placebo group

SUMMARY:
The purpose of the present study was to evaluate the effects of subgingival delivery of 1.2% Rosuvastatin (RSV) gel as an adjunct to scaling and root planing in chronic periodontitis (CP) with Type 2 diabetes mellitus patients.

DETAILED DESCRIPTION:
Background: The purpose of this double-masked, randomized, controlled clinical trial was to evaluate the effects of subgingival delivery of 1.2% Rosuvastatin gel as an adjunct to scaling and root planing (SRP) on clinical and radiographic parameters and compare this method with SRP plus placebo gel alone in chronic periodontitis (CP) with type 2 DM patients.

Methods: Eighty CP patients with type 2 DM are included in this study. They were divided into two groups: 1) SRP + 1.2% Rosuvastatin gel (RSV group); 2) SRP + Placebo gel (Placebo group). At baseline, 3, 6 and 9 months after treatment, clinical measurements, including plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), clinical attachment level (CAL) and radiographic parameters intrabony defect depth (IBD), percentage change in radiographic defect depth reduction (DDR%) were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with deep pockets (PD of ≥5mm or CAL ≥4mm) and vertical bone loss ≥3 mm on intraoral periapical radiographs
* Patients with ≥20 teeth with no history of periodontal therapy in the preceding 6 months nor under any antibiotic therapy

Exclusion Criteria:

* Patients with any other known systemic disease
* Patients on systemic statin therapy
* Known or suspected allergy to statin supplementation
* Patients with aggressive periodontitis
* Tobacco use in any form, smokers, alcoholics
* Immunocompromised patients
* Pregnant or lactating females

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Defect depth reduction (%) | Change from baseline to 9 months
  Assessed in percentage

SECONDARY OUTCOMES:
probing depth (mm) | Change from baseline to 9 months
  measured in mm
clinical attachment level (mm) | Change from baseline to 9 months
  measured in mm
modified sulcus bleeding index | Change from baseline to 9 months
  scale from 0-3
plaque index | Change from baseline to 9 months
  scale from 0-3

CONTACTS AND LOCATIONS:
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India